CLINICAL TRIAL: NCT00265642
Title: Study of the Effects of a Sartan on Hepatic Fibrosis Progression in Chronic Viral Hepatitis C
Brief Title: Evaluation of Irbesartan on Hepatic Fibrosis in Chronic Hepatitis C
Acronym: Fibrosar
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-006027-37; ANRS HC 19 Fibrosar
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2012-07

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; irbesartan
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group verum (Experimental): Drug: Irbesartan
  Interventions: Drug: Irbesartan
- group placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Irbesartan — one tablet of 150 mg/d during 2 years
  Arms: group verum
Drug: placebo — one tablet per day during 2 years
  Arms: group placebo

SUMMARY:
The purpose of this study is to examine the efficacy of irbesartan on the progression of liver fibrosis in adult patients with chronic hepatitis C.

The expected total enrollment is 200 patients. Patients who meet the study criteria and accept to participate at this study will take by day one tablet of 150 mg of treatment (irbesartan or placebo) during two years. The assessment of efficacy will be make by evaluation of area of liver fibrosis and blood markers of liver fibrosis

DETAILED DESCRIPTION:
The results of several studies suggests than the AT1 receptor antagonists of angiotensin II have inhibitory effects on TGF-beta 1 production and can limit the progression of liver fibrosis.

Therefore, the angiotensin II could be another mediator of the synthesis of the extra-cellular matrix at the hepatic level, opening new perspectives with the antagonists of angiotensin II receptors drugs (ARA2/sartans).

This study is a randomized, double blind, multi-center, parallel assignment, and efficacy study.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* liver biopsy performed (less 18 month before inclusion), fibrosis score F2,F3 or F3+ in Metavir classification,
* patients without antiviral therapy
* contraindication to anti viral treatment
* non responders or relapsers patients to past antiviral treatment

Exclusion Criteria:

* hepatocellular carcinoma
* HIV
* alcool abuser
* cirrhosis
* anti-fibrotic treatment
* pregnancy or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2006-10; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Assessment of liver fibrosis changes by measurement of area of porto-septal fibrosis (morphometry)at M24 | at M24

SECONDARY OUTCOMES:
Assessment of liver fibrosis changes at M24 by non-invasive tests ((blood test mainly and also elastometry) | at M24

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cales, MD, Principal Investigator — CHU Angers, Service d'hépato-gastroentérologie, 49933 Angers Cedex 09; Fabrice Carrat, MD, Study Chair — Inserm U707 France
Locations (1):
- CHU Angers, Service d'hépato-gastroentérologie, Angers, France

REFERENCES:
- See also: Related Info — http://www.anrs.fr